CLINICAL TRIAL: NCT05919160
Title: Assessment of Safety and Utility of a High-density Microelectrode for Human Neuronal Recording
Brief Title: A High-density Microelectrode for Human Neuronal Recordings
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Adam Mamelak, MD, Professor of Neurosurgery, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: STUDY00002777
Record Dates: First submitted 2023-06-09; First posted 2023-06-26 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Parkinson Disease, Idiopathic
Keywords: Parkinson's; DBS; Electrode
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Neuronal Recording and Behavioral Testing (Experimental): Neuronal Recording and Behavioral Testing
  Interventions: Device: DBC (Diagnostic Biochips) Deep Array microelectrode; Intan Electrophysiology recording system; Matlab response recording to behavioral task

INTERVENTIONS:
Device: DBC (Diagnostic Biochips) Deep Array microelectrode; Intan Electrophysiology recording system; Matlab response recording to behavioral task — Devices listed are components of a single intervention that includes: Record neuronal activity (Intan) from electrodes (DBC), record and analyze patient responses (Matlab)

SUMMARY:
The purpose of this study is to test the ability of a newly-designed electrode to measure the activity of individual nerve cells (neurons), and collections of nerve cells (local field potentials) in the brain. The study's main goals are to see how well this electrode works compared to standard electrodes and to validate its safety.

DETAILED DESCRIPTION:
Recording of human brain activity at many scales is an important tool in clinical medicine. The ability to record extracellular action potentials, otherwise known as a "single unit activity" (SUA) has provided fundamental insight into the details of neuronal function in humans as well as a variety of nonhuman animals. In humans the techniques for recording extracellular action potentials are relatively limited. Rigid, sharp tipped probes manufactured by several companies are FDA approved and routinely used as part of standard of care during a variety of surgical procedures such as deep brain stimulation (DBS) device implantation to identify areas of neuronal activity and optimize placement of clinical electrodes. The same technique has been used to better understand brain function and its impairment by disease in humans. In addition, a variety of semi- chronically implanted microwire techniques are available. These electrodes are more commonly used in patients with seizure disorders and have allowed insight into network behavior such as in the medial temporal lobe and medial frontal lobe.

However there remains a tremendous gap between the recording capabilities of modern electrodes used in animal research, and what is currently clinically available for human testing. A typical rigid shaft single electrode currently used in clinical care will record anywhere from 1-3 distinctly isolated neurons at a time. In contrast, in state-of-the art animal research, higher density probes such as the Neuropixel electrode [4-6] now routinely allow recording of hundreds or even thousands of neurons in a single brain region. This markedly increased recording capability translates directly into a better understanding of how brain neurons and networks interact to create complex behaviors and disease. Most of the commonly used high-density electrodes are based on a rigid silicon shaft onto which multiple recording contacts (typically made of platinum, Iridium, gold or conductive polymers) are embedded. There are several significant limitations of silicon-based probes in translating them to large brain, and in particular human, applications [7] First, silicon is fragile, making the electrodes prone to fracture, which makes them risky for human applications. Furthermore, the silicon microfabrication process is impractical for making large devices, limiting commercially available probe length to around 20mm, which is too short for most clinical applications in the human brain. Also, the connection between the electrode contacts and the pre-amplifier in the currently available products requires a rigid circuit board that is attached to the electrode, which is difficult to work with and which requires that the pre-amplifiers to be kept very close to the brain. While there are FDA approved version of silicon probes (i.e. the Utah Array used for brain machine interfaces), these applications are limited to short <2mm long probes used for surface cortical recordings. The inherent material and process limitations described make it unlikely that silicon-based probe technologies will provide a clinically usable probe for deeper locations in the human brain. The investigators, therefore, sought to utilize a new kind of translatable technology for clinical use.

The investigators seek to test a more robust and reliable technique for recording large numbers of single neurons in the human brain. Diagnostic Biochips Inc. (Glen Burnie, MD) is an electrode manufacturer that has developed a new type of electrode that consists of a stainless-steel shaft and an array of polyimide based high density electrodes that are embedded onto this shaft. This type of electrode design has proven highly reliable for deep brain penetrations of up to of up to 8cm length in rodent and non-human primate. The steel carrier is highly robust, entirely avoiding the breakage problems associated with silicon based and other high-density probe designs. Similarly, the polyimide-based electrodes are a material that is well known to not be biotoxic, which is well tolerated and part of numerous currently FDA approved products. The DBC Deep Array electrode is wired directly to an Intan (Los Angeles, CA) microprocessor mounted at the other end of the shaft. This microprocessor generates a digital signal, so that a long connection can be utilized between the microprocessor and Intan amplifier unit used to record the data, without any loss in signal or addition of noise. This feature is crucial to improve patient safety and reduce any infection risks during recording. Steel is rigid, and not prone to fracture like silicon. In addition, this type of electrode can be made significantly longer, simply by using a longer stainless-steel shaft to mount the high-density polyimide array on. While the currently manufactured DBC deep arrays used in animal research are 40-80 mm in length, a length of up to 300 mm is easily feasible. This contrasts with the maximal 10 -20 mm length that is achievable for silicon-based and other high-density systems. A length of >100mm is required for probing deep brain structures such as the basal ganglia in the human brain, which is routinely done in clinical settings. The DBC electrode can record up to 1024 individual channels simultaneously. The DBC devices have been used successfully in nonhuman primates and have undergone the biocompatibility, cytotoxicity, sterilization, and safety testing expected for use in humans. The results of these tests were all a pass, and the resulting reports are attached to this protocol.

ELIGIBILITY:
Inclusion Criteria:

* Any patient undergoing implantation of a Deep Brain Stimulating (DBS) electrode in the Subthalamic nucleus (STN) for the treatment of Parkinson's disease, in whom microelectrode recording is being performed to improve localization of the STN.
* Age > 18 years of age
* Able to give independent informed consent

Exclusion Criteria:

* Microelectrode recording is not indicated
* Previous implantation of DBS electrodes in this site
* Known allergic reaction to stainless steel or polyimide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Neuronal Activity | One week after recording in OR completed
  Single Neuron firing rate (spikes) measured in spikes per second - total number of isolated neurons, amplitude (in uV of spikes) - by Intan Neurophysiology Recording System
Breakage of Electrode | One week after recording in OR completed
  Extent of fracture of electrode tip measured in micrometers by a light microscope

CONTACTS AND LOCATIONS:
Overall Officials: Adam Mamelak, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No